CLINICAL TRIAL: NCT01503892
Title: Metanx Effects on Nerve Fiber Density in Neuropathic Diabetics
Acronym: SLHN2011-18
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Collaborators: Goldfarb Foundation (Unknown); Pamlab, L.L.C. (Industry)
Responsible Party: Principal Investigator, Edwin S. Hart III, Principal Investigator, St. Luke's Hospital and Health Network, Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: StLukeHHN
Record Dates: First submitted 2011-12-29; First posted 2012-01-04 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes; Peripheral Neuropathy
Keywords: Small Fiber Neuropathy; Metanx Effect on Small Fiber Neuropathy; Metanx Effect on Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases; Small Fiber Neuropathy | interventions — metanx

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The control group will receive placebo pill twice daily for twelve months.
  Interventions: Drug: Placebo
- Metanx (Active Comparator): Metanx group will receive one pill twice daily for twelve months.
  Interventions: Dietary Supplement: Metanx

INTERVENTIONS:
Dietary Supplement: Metanx — Metanx- one tablet twice daily for twelve months
  Arms: Metanx
Drug: Placebo — Placebo- one tablet twice daily for twelve months.
  Arms: Placebo

SUMMARY:
This study focuses on the use of Metanx® as the sole treatment for improving and reversing nerve damage in type 2 diabetic patients with peripheral neuropathy. There will be two equal study groups enrolled in this randomized double blinded study. The minimum sample size of enrollment is 24 (12 per group), which is required for 90% power at alpha = .05. The maximum number of participants will be set at 100 (50 per group). Patients who are pre-diabetic or patients who have been diagnosed with diabetes type II for less than five years are included in this study. The control group will receive placebo pill twice daily versus the treatment group which will receive one Metanx® tablet twice daily. Each group will have intraepidermal nerve fiber densities obtained by skin biopsies taken at the beginning of the study before any treatment has begun as well as a final intraepidermal nerve skin biopsy at the end of twelve months to re-biopsy. In addition each group will answer three sets of questionnaires relating to their peripheral neuropathy at initial, three months, twelve month visitations. If Metanx® is able to reverse nerve damage and improve symptoms then the final nerve biopsies will show an increase in intraepidermal nerve fiber density and an improvement in the subjective score versus the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetics
* Pre-diabetics
* Symptoms of peripheral neuropathy

Exclusion Criteria:

* Pregnancy
* Under age 18
* HIV (+)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Increased intraepidermal nerve fiber density | 1 year
  If Metanx® is able to reverse nerve damage and improve symptoms then the final nerve biopsies will show an increase in intraepidermal nerve fiber density

SECONDARY OUTCOMES:
Subjective improvement | 1 year
  Improvement in the subjective score versus the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin S. Hart III, DPM, Principal Investigator — St. Luke's Hospital and Health Network
Locations (1):
- St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania, United States

REFERENCES:
- See also: William L. Goldfarb Educational Foundation for Research and Teaching of the Lower Extremity — http://www.goldfarbfoundation.org/
- See also: St. Luke's Hospital and Health Network — http://www.mystlukesonline.org